CLINICAL TRIAL: NCT03778346
Title: Integrin β7, BCMA, CS1, CD38 and CD138 as the Single or Compound Targets for the Fourth Genenation of CAR-T Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Sixth Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Zhejiang Qixin Biotech (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SixthAHWenzhouMU
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: RRMM
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T therapy in multiple myeloma (Experimental): In order to assess the safety and validity of using the Fourth Genenation of CAR-T therapy refractory/rela-psed multiple myeloma patients with one kind of BCMA-CART,CD138-CART,CD38-CART , Integrin β7-CART or 10 different combinations ,subjects will receive 10^6-10^7/Kg transduced CAR-T cells at one time.
  Interventions: Biological: CAR-T therapy in Relapsed/Refractory multiple myeloma

INTERVENTIONS:
Biological: CAR-T therapy in Relapsed/Refractory multiple myeloma — Integrin β7, BCMA, CS1, CD38 and CD138 as the Single or Compound Targets for the Fourth Genenation of CAR-T Cells to treat Relapsed/Refractory multiple myeloma

SUMMARY:
According to the high expression of tumor cell-associated antigen CD138, integrin β7, CS1, CD38 and BCMA in patients with refractory/recurrent multiple myeloma, the fourth generation of CAR-T cells(simultaneously expressing IL7 and CCL19) with 10 different dual target combinations are used to minimize the tumor burden in the patient individually and precisely and improve the immunosuppressive microenvironment of the tumor , thereby effectively treating refractory/recurrent multiple myeloma .

DETAILED DESCRIPTION:
Multiple myeloma（MM） is one of the most common malignant diseases in the blood system.There is still no cure for the disease which only control the development of the disease in various ways including proteasome inhibitors and immune regulator and hematopoietic stem cell transplantation . Combined with the advantages of multiple therapies, chimeric antigen receptor T cells (CAR-T) have gradually becoming one of the strongest and most powerful weapons against multiple myeloma.The basic principle is to use the patient's own immune cells to clear cancer cells.

MM is genetically and phenotypically heterogeneous,Antigen escape and relapse after CAR-T treatment is a global problem， so the effective treatment of refractory/relapsing multiple myeloma with CAR-T cells usually requires targeting multiple antigens. The investigators use Integrin β7(a large family of molecules that are central regulators in multicellular biology and orchestrating cell-cell and cell-extracellular matrix (ECM) adhesive interactions from embryonic development to mature tissue function), BCMA(highly expressed on malignant MM plasma cells and providing a substantial antiapoptotic signal making it an encouraging target for BCMA-directed immunotherapy),CS1(encoded by the SLAMF7 gene,a robust marker of normal plasma cells and malignant plasma),CD38(encoded by the CD38 gene and functioning in cell adhesion, signal transduction and calcium signaling) and CD138(known as syndecan 1, a surface protein expressed on most healthy and malignant plasma cells as an adhesion protein, binding collagen and fibronectin molecules located in the extracellular matrix. ) as the Single or Compound Targets for the Fourth Genenation of CAR-T Cells ,thereby effectively treating refractory/recurrent multiple myeloma .

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the requirements voluntarily participate in the study and sign the Informed Consent Form.
2. Age is 18 to 80 years old, gender is not limited.
3. Patients with relapsed or refractory myeloma who meet the following criteria for multiple myeloma diagnostic criteria defined by the IMWG (2017): Subjects have received adequate prior treatment of at least 2 regimens; during the most recent treatment or after treatment , the disease progresses or recurs.
4. The Eastern Cancer Cooperative Group (ECOG) scores 0 to 2 (the tumor causes bone pain).
5. The expected survival period is more than 12 weeks.
6. No other malignant tumors, severe autoimmune diseases or congenital immunodeficiency, serious progressive infection, cranial nerve disorder or mental illness.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with uncontrollable active infections.
3. Patients with systemic steroids; recent or current use of inhaled steroids is not excluded.
4. Previously involved CAR-T cell therapies produced any uncontrolled disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events that are related to treatment | 2 years
  Safety and tolerability measured by occurrence of study related adverse effects defined by NCI-CTCAE v4.03

SECONDARY OUTCOMES:
2 year overall survival(OS) | 2 yaers
  To estimate 2 year overall survival(OS) after BCMA/CD138/CD38/Integrinβ7/CS1-CART infusion and sequential treatment with Relapsed/Refractory MM
3 year progression free survival (PFS) | 3 yaers
  To estimate 3 year progression free survival after BCMA/CD138/CD38/Integrinβ7/CS1 CART infusion and sequential treatment with Relapsed/Refractory MM

CONTACTS AND LOCATIONS:
Overall Officials: Bingmu Fang, M.D, Principal Investigator — Lishui Country People's Hospital
Locations (3):
- China (3):
  - Jinhong Jiang, Lishui, Zhejiang
  - The Sixth Affiliated Hospital of Wenzhou Medical University, Lishui, Zhejiang
  - Zhejiang QiXin Biotech, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruella M, Barrett DM, Kenderian SS, Shestova O, Hofmann TJ, Perazzelli J, Klichinsky M, Aikawa V, Nazimuddin F, Kozlowski M, Scholler J, Lacey SF, Melenhorst JJ, Morrissette JJ, Christian DA, Hunter CA, Kalos M, Porter DL, June CH, Grupp SA, Gill S. Dual CD19 and CD123 targeting prevents antigen-loss relapses after CD19-directed immunotherapies. J Clin Invest. 2016 Oct 3;126(10):3814-3826. doi: 10.1172/JCI87366. Epub 2016 Aug 29. PMID 27571406
- [Background] Adachi K, Kano Y, Nagai T, Okuyama N, Sakoda Y, Tamada K. IL-7 and CCL19 expression in CAR-T cells improves immune cell infiltration and CAR-T cell survival in the tumor. Nat Biotechnol. 2018 Apr;36(4):346-351. doi: 10.1038/nbt.4086. Epub 2018 Mar 5. PMID 29505028
- [Background] Petrov JC, Wada M, Pinz KG, Yan LE, Chen KH, Shuai X, Liu H, Chen X, Leung LH, Salman H, Hagag N, Liu F, Jiang X, Ma Y. Compound CAR T-cells as a double-pronged approach for treating acute myeloid leukemia. Leukemia. 2018 Jun;32(6):1317-1326. doi: 10.1038/s41375-018-0075-3. Epub 2018 Feb 25. PMID 29515236
- [Background] Lim WA, June CH. The Principles of Engineering Immune Cells to Treat Cancer. Cell. 2017 Feb 9;168(4):724-740. doi: 10.1016/j.cell.2017.01.016. PMID 28187291
- [Background] Hosen N, Matsunaga Y, Hasegawa K, Matsuno H, Nakamura Y, Makita M, Watanabe K, Yoshida M, Satoh K, Morimoto S, Fujiki F, Nakajima H, Nakata J, Nishida S, Tsuboi A, Oka Y, Manabe M, Ichihara H, Aoyama Y, Mugitani A, Nakao T, Hino M, Uchibori R, Ozawa K, Baba Y, Terakura S, Wada N, Morii E, Nishimura J, Takeda K, Oji Y, Sugiyama H, Takagi J, Kumanogoh A. The activated conformation of integrin beta7 is a novel multiple myeloma-specific target for CAR T cell therapy. Nat Med. 2017 Dec;23(12):1436-1443. doi: 10.1038/nm.4431. Epub 2017 Nov 6. PMID 29106400
- [Background] Drent E, Groen RW, Noort WA, Themeli M, Lammerts van Bueren JJ, Parren PW, Kuball J, Sebestyen Z, Yuan H, de Bruijn J, van de Donk NW, Martens AC, Lokhorst HM, Mutis T. Pre-clinical evaluation of CD38 chimeric antigen receptor engineered T cells for the treatment of multiple myeloma. Haematologica. 2016 May;101(5):616-25. doi: 10.3324/haematol.2015.137620. Epub 2016 Feb 8. PMID 26858358
- [Background] Brudno JN, Maric I, Hartman SD, Rose JJ, Wang M, Lam N, Stetler-Stevenson M, Salem D, Yuan C, Pavletic S, Kanakry JA, Ali SA, Mikkilineni L, Feldman SA, Stroncek DF, Hansen BG, Lawrence J, Patel R, Hakim F, Gress RE, Kochenderfer JN. T Cells Genetically Modified to Express an Anti-B-Cell Maturation Antigen Chimeric Antigen Receptor Cause Remissions of Poor-Prognosis Relapsed Multiple Myeloma. J Clin Oncol. 2018 Aug 1;36(22):2267-2280. doi: 10.1200/JCO.2018.77.8084. Epub 2018 May 29. PMID 29812997
- [Background] Bu DX, Singh R, Choi EE, Ruella M, Nunez-Cruz S, Mansfield KG, Bennett P, Barton N, Wu Q, Zhang J, Wang Y, Wei L, Cogan S, Ezell T, Joshi S, Latimer KJ, Granda B, Tschantz WR, Young RM, Huet HA, Richardson CJ, Milone MC. Pre-clinical validation of B cell maturation antigen (BCMA) as a target for T cell immunotherapy of multiple myeloma. Oncotarget. 2018 May 25;9(40):25764-25780. doi: 10.18632/oncotarget.25359. eCollection 2018 May 25. PMID 29899820
- [Background] Mikkilineni L, Kochenderfer JN. Chimeric antigen receptor T-cell therapies for multiple myeloma. Blood. 2017 Dec 14;130(24):2594-2602. doi: 10.1182/blood-2017-06-793869. Epub 2017 Sep 19. PMID 28928126
- [Background] Chmielewski M, Abken H. TRUCKs: the fourth generation of CARs. Expert Opin Biol Ther. 2015;15(8):1145-54. doi: 10.1517/14712598.2015.1046430. Epub 2015 May 18. PMID 25985798
- [Derived] Duan D, Wang K, Wei C, Feng D, Liu Y, He Q, Xu X, Wang C, Zhao S, Lv L, Long J, Lin D, Zhao A, Fang B, Jiang J, Tang S, Gao J. The BCMA-Targeted Fourth-Generation CAR-T Cells Secreting IL-7 and CCL19 for Therapy of Refractory/Recurrent Multiple Myeloma. Front Immunol. 2021 Mar 5;12:609421. doi: 10.3389/fimmu.2021.609421. eCollection 2021. PMID 33767695